CLINICAL TRIAL: NCT04246671
Title: Phase 1 Trial of Intravenous Administration of TAEK-VAC-HerBy Vaccine Alone and in Combination With HER2 Antibodies in Patients With Advanced Cancer.
Brief Title: TAEK-VAC-HerBy Vaccine for Brachyury and HER2 Expressing Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAEK-VAC-HerBy-001
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Chordoma; HER2-positive Breast Cancer
Keywords: Brachyury; HER2-expessing cancer
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Stage 1 dose escalation: TAEK-VAC-HerBy (1x10E7 Inf.U) (Experimental): TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose level 1x10E7 Inf.U.
  Interventions: Biological: TAEK-VAC-HerBy
- Stage 1 dose escalation: TAEK-VAC-HerBy (1x10E8 Inf.U) (Experimental): TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose level 1x10E8 Inf.U.
  Interventions: Biological: TAEK-VAC-HerBy
- Stage 1 dose escalation: TAEK-VAC-HerBy (1x10E9 Inf.U) (Experimental): TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose level 1x10E9 Inf.U.
  Interventions: Biological: TAEK-VAC-HerBy
- Stage 1 dose escalation: TAEK-VAC-HerBy (1x10E10 Inf.U) (Experimental): TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose level 1x10E10 Inf.U.
  Interventions: Biological: TAEK-VAC-HerBy
- Stage 2: Chordoma Cancer Cohort (Experimental): TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose level defined in stage 1.
  Interventions: Biological: TAEK-VAC-HerBy
- Stage 2: HER2-positive Breast Cancer Cohort (Trastuzumab + TAEK-VAC-HerBy) (Experimental): TAEK-VAC-HerBy will be administered intravenously to patients who are on stable dose of trastuzumab, every three weeks with three administrations in total at the dose defined in stage 1.
  Interventions: Biological: TAEK-VAC-HerBy

INTERVENTIONS:
Biological: TAEK-VAC-HerBy — TAEK-VAC-HerBy will be administered intravenously every three weeks with three administrations in total at the dose defined in stage 1. During stage 2, it may also be administered concurrently with a HER2 antibody(ies) (trastuzumab, pertuzumab).

SUMMARY:
A Phase 1 open label trial of intravenous administration of TAEK-VAC-HerBy vaccine in patients with advanced brachyury and/or HER2- expressing cancer. The study will be completed in 2 stages. In Stage 1 patients will be enrolled and treated according to a 3+3 dose escalation scheme. Up to 4 dose levels will be explored to determine the recommended dose of TAEK-VAC-HerBy for Stage 2 of the trial. Stage 2 will enroll either chordoma patients for treatment with TAEK-VAC-HerBy alone, or HER2- positive breast cancer patients for combination treatment of TAEK-VAC-HerBy vaccine and therapeutic HER2 antibodies (trastuzumab). Patients in both stages will receive TAEK-VAC-HerBy intravenously, every three weeks, three administrations in total.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria, apply to all cohorts:

* Men and women ≥18 years old.
* Patients must have histologically documented malignant tumor which is unresectable locally advanced or metastatic.
* ECOG performance status 0 or 1
* Patients must have normal organ and bone marrow function as defined in the protocol.
* Normal left ventricular ejection fraction (LVEF) ≥50%.
* Troponin I within normal limits.
* A maximum cumulative dose of prior doxorubicin ≤360 mg/m2 or epirubicin ≤720 mg/m2
* Any approved cancer therapy (except HER2 antibodies) must be completed at least 3 weeks or 5 half-lives for small molecule inhibitors, whichever is shorter, prior to the first planned dose of TVH vaccine.
* HER-2 positive cancer: Patients are required to be on active treatment with HER2 antibodies (trastuzumab) prior to and during study treatment.
* Chordoma patients with progressive extracranial chordoma (base of skull is permitted) not amenable for surgical resection with curative intent, nor for radiation therapy will be enrolled.
* Patients must have recovered (Grade 1 or baseline) from any clinically significant toxicity associated with prior therapy.
* Patients must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1.

Exclusion Criteria:

* Known metastatic disease to the central nervous system, unless previously treated and responded with a minimum stable disease over 2 CT scans separated at least 4 weeks from each other, and more than 6 weeks since the last dose of dexamethasone.
* History of allergy or untoward reaction to prior vaccination with vaccinia virus, aminoglycoside antibiotics, ciprofloxacin, or egg products.
* Subjects should have no known evidence of being immunocompromised.
* Chronic administration (defined as >5 consecutive days of >15 mg of prednisone (or equivalent) per day) of systemic corticosteroids within 14 days of the first planned dose of TAEK-VAC-HerBy vaccine. Use of inhaled steroids, nasal sprays, eye drops, and topical creams is allowed. Steroids premedication for CT scans is allowed.
* Clinically significant cardiomyopathy, coronary disease, congestive heart failure (NYHA class III or IV) or reduced as per institutional standards LVEF, poorly controlled hypertension (systolic >180 mm Hg or diastolic >100 mm Hg) or cerebrovascular accident within 1 year.
* Known history of, or any evidence of active, non-infectious pneumonitis or primary pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Patients with Dose Limiting Toxicity (DLT) | DLT evaluation period is 30 days after the last vaccine dose
  Frequency of patients with DLTs

CONTACTS AND LOCATIONS:
Overall Officials: Mary (Nora) L Disis, MD, Principal Investigator — University of Washington Medicine Seattle
Locations (9):
- United States (9):
  - Mayo Clinic - Phoenix, Scottsdale, Arizona
  - Providence Saint John's Health Center, Santa Monica, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Center Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Providence Cancer Institute, Portland, Oregon
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694